CLINICAL TRIAL: NCT05322980
Title: Microcephaly At Birth As a Potential Predictor of Poor Prognosis in Infants Weighing 500 Grams or Less: a Retrospective Cohort Study
Brief Title: Summary of Infants Weighing 500 Grams or Less
Status: Completed | Type: Observational
Sponsor: Nagano Children's Hospital (Other)
Responsible Party: Principal Investigator, Ryo Itoshima, Researcher, Nagano Children's Hospital
Other Study IDs: summary-500g
Record Dates: First submitted 2022-03-04; First posted 2022-04-12 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Infant, Extremely Low Birth Weight; Microcephaly
Keywords: 500 grams or less; prognosis
MeSH Terms: conditions — Microcephaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Microcephaly: Infants with primary microcephaly.
  Interventions: Diagnostic Test: Microcephaly
- Control: Infants without primary microcephaly.

INTERVENTIONS:
Diagnostic Test: Microcephaly — Those with a z score of birth head circumference < -2 (primary microcephaly) are classified into the Microcephaly group.
  Groups: Microcephaly

SUMMARY:
This is a retrospective single-center cohort study. The comparison in short- and long-term outcomes will be made between those with and without primary microcephaly in infants weighing ≤ 500 g.

DETAILED DESCRIPTION:
This is a retrospective single-center cohort study. The study setting is a level IV neonatal intensive care unit (NICU) at Nagano Children's Hospital in Nagano, Japan. We will retrospectively collect the data of those who were admitted to Nagano Children's Hospital NICU between January 1, 2015, and December 31, 2019. Eligible infants will be identified using our neonatal database and clinical records. The extracted data includes maternal background information and clinical course, infant's status at birth, the clinical course in NICU, and the follow-up data at 6 and 18 months of corrected age.

Among the eligible infants, those with a z score of birth head circumference < -2 will be classified into the Microcephaly group and others into the Control group. The z score is calculated using the Japanese growth standard.

ELIGIBILITY:
Inclusion Criteria:

* Live-born infants weighing ≤ 500 g at birth
* Infants whose clinical course is available in the electronic medical record

Exclusion Criteria:

* Stillbirths
* Infants who received only palliative care at birth
* Outborn infants
* Infants whose assessment at 3 years of age not completed at data analysis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Those who were admitted to Nagano Children's Hospital NICU between January 1, 2010, and December 31, 2019.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of neurodevelopmental impairment | 3 years of age
  Having at least one of the following conditions: cognitive impairment, cerebral palsy, visual impairment, or hearing impairment. Cognitive impairment was defined as a modified DQ score of ≤ 70 using the Kyoto Scale of Psychological Development. CP was defined as (1) a non-progressive disorder of the central nervous system appearing in the early years of life and clinically characterized by a persistent but not unchanging impairment of movement and posture and/or (2) the Gross Motor Function Classification System level ≥ II. Visual impairment was defined as unilateral or bilateral blindness, or any other condition requiring corrective lenses, which were diagnosed or determined by ophthalmologists. Hearing impairment was defined as unilateral or bilateral hearing loss that requires a hearing aid. The diagnosis of hearing loss was made by otolaryngologists using auditory steady-state response.

SECONDARY OUTCOMES:
Survival rate | At discharge from neonatal intensive care unit, an average at 40 weeks' postmenstrual age.
  Survival rate is the proportion of those have survived.
Rate of severe bronchopulmonary dysplasia | At 36 weeks' postmenstrual age
  The definition of bronchopulmonary dysplasia proposed by the National Institute of Child Health and Human Development is used to classify the severity of bronchopulmonary dysplasia. Those who need ≥ 30% of oxygen or any mechanical respiratory support at 36 weeks of gestation are classified as having severe bronchopulmonary dysplasia.
Rate of need for surgery for patent ductus arteriosus | In neonatal intensive care unit, an average of up to 4 weeks of life
  Patent ductus arteriosus is diagnosed by neonatologists using echocardiography and clinical signs.
Rate of severe intraventricular hemorrhage | In neonatal intensive care unit, an average of up to 2 weeks of life
  Intraventricular hemorrhage is diagnosed by neonatologists using head ultrasound. Severe IVH was defined as grade III or IV by the classification of Papile.
Rate of periventricular leukomalacia | In neonatal intensive care unit, an average of up to 40 weeks' postmenstrual age
  Periventricular leukomalacia is diagnosed using head ultrasound or magnetic resonance imaging, typically cysts formation in the periventricular white matter.
Rate of necrotizing enterocolitis | In neonatal intensive care unit, an average of up to 2 weeks of life
  The diagnosis with necrotizing enterocolitis.
Rate of sepsis | In neonatal intensive care unit, an average of up to 4 weeks of life
  Sepsis is defined as septicemia or bacteremia with a positive culture result of the blood and/or cerebrospinal fluid.
Rate of need for treatment for retinopathy of prematurity | In neonatal intensive care unit, an average of up to 40 weeks' postmenstrual age
  The diagnosis of retinopathy of prematurity and the decision on the need for treatment were made by ophthalmologic examination.
Weight | At 40 weeks' postmenstrual age or at discharge (approximately 40 weeks' postmenstrual age)
  Physical measurement.
Length | At 40 weeks' postmenstrual age or at discharge (approximately 40 weeks' postmenstrual age)
  Physical measurement.
Head circumference | At 40 weeks' postmenstrual age or at discharge (approximately 40 weeks' postmenstrual age)
  Physical measurement.
Postmenstrual age | At discharge, an average at 40 weeks' postmenstrual age
  Postmenstrual age is calculated based on their gestational age and date at birth.
Need for home oxygen therapy | At discharge, an average at 40 weeks' postmenstrual age
  Need for home oxygen therapy.
Tracheostomy | In neonatal intensive care unit, an average at 40 weeks' postmenstrual age
  Need for tracheostomy.
Length of hospital stay | In neonatal intensive care unit, an average at 40 weeks' postmenstrual age
  The initial hospitalization.
Survival rate | At 3 years of age
  Survival rate is the proportion of those have survived.
Modified developmental quotient | At 3 years of age
  Modified developmental quotient is calculated by dividing developmental age (measured by the Kyoto Scale of Psychological Development) by the corrected age.
Rate of cerebral palsy | At 3 years of age
  Cerebral palsy is defined as (1) a non-progressive disorder of the central nervous system appearing in early years of life and clinically characterized by a persistent but not unchanging impairment of movement and posture and/or (2) the Gross Motor Function Classification System level ≥ II.
Rate of visual impairment | At 3 years of age
  Visual impairment is defined as unilateral or bilateral blindness, or any other condition requiring corrective lenses, which were diagnosed or determined by ophthalmologists.
Rate of hearing impairment | At 3 years of age
  Hearing impairment is defined as unilateral or bilateral hearing loss that requires a hearing aid. The diagnosis of hearing loss was made by otolaryngologists using auditory steady-state response.
Rate of those who need home oxygen therapy | At 3 years of age
  Need for home oxygen therapy.
Rate of those who need tracheostomy | At 3 years of age
  Need for tracheostomy.
Rate of those who need tube feeding or gastrostomy | At 3 years of age
  Need for tube feeding or gastrostomy.
Rate of those who need rehospitalization | After 18 months of corrected age unit until 3 years of age
  Need for rehospitalization.
Weight | At 3 years of age
  Physical measurement.
Height | At 3 years of age
  Physical measurement.
Head circumference | At 3 years of age
  Physical measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Ryo Itoshima, MD, Principal Investigator — Nagano Children's Hospital
Locations (1):
- Nagano Children's Hospital, Azumino, Nagano, Japan

IPD SHARING:
Plan to Share IPD: No